CLINICAL TRIAL: NCT06958029
Title: Incidence and Risk Factors of Postoperative Atrial Fibrillation in Cardiac Surgery Patients
Brief Title: Postoperative Atrial Fibrillation in Cardiac Surgery
Acronym: POAF
Status: Recruiting | Type: Observational
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Thepakorn Sathitkarnmanee, Associate professor, Khon Kaen University
Other Study IDs: HE671492; Khon Kaen University (Other: Khon Kaen University)
Record Dates: First submitted 2025-04-27; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Post-operative Atrial Fibrillation
Keywords: postoperative; atrial fibrillation; cardiac surgery
MeSH Terms: conditions — Atrial Fibrillation | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac surgery: Patients undergoing cardiac surgery
  Interventions: Procedure: Cardiac surgery

INTERVENTIONS:
Procedure: Cardiac surgery — Patients receiving general anesthesia for cardiac surgery

SUMMARY:
This multicenter observational study aims to investigate the incidence and identify risk factors associated with postoperative atrial fibrillation (POAF) in patients undergoing cardiac surgery at three medical centers in Thailand. The study will examine patient characteristics, surgical factors, and anesthetic management practices that may contribute to the development of this common postoperative complication.

DETAILED DESCRIPTION:
Postoperative atrial fibrillation (POAF) is a common complication following cardiac surgery, with incidence rates reported between 15-30% after valve surgery and 18-74% after coronary artery bypass grafting. POAF typically occurs within 72 hours after surgery and is associated with increased morbidity, mortality, length of hospital stay, and healthcare costs.

The Society of Thoracic Surgeons has identified five major postoperative complications associated with cardiac surgery, including POAF, which can significantly affect patient outcomes. This multicenter observational study will examine the incidence and risk factors of POAF in cardiac surgery patients across three medical centers in Thailand: Srinagarind Hospital at Khon Kaen University, Northeastern Thailand Cardiac Center, and Surat Thani Hospital.

The study will collect data on patient demographics, comorbidities, preoperative laboratory values, perioperative characteristics, surgical procedures (valve surgery, CABG, combined procedures), and postoperative complications. By identifying risk factors associated with POAF, this study aims to develop preventive strategies and improve management protocols for patients at high risk for this complication.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients undergoing cardiac valve surgery or coronary artery bypass grafting (CABG) procedures

Exclusion Criteria:

* Patients undergoing aortic surgery
* Patients undergoing MAZE procedure
* Incomplete medical records
* Patients who required mechanical circulatory support before surgery
* Patients who died during surgery or within 3 days after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ubdergoing cardiac surgery
Sampling Method: Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Incidence | 72 hours postoperatively
  The incidence of POAF

SECONDARY OUTCOMES:
Risk factors | 72 hours postoperatively
  Risk factors associated with POAF

CONTACTS AND LOCATIONS:
Overall Officials: Thepakorn Sathitkarnmanee, MD, Principal Investigator — Khon Kaen University
Locations (1):
- Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand

REFERENCES:
- [Result] Crawford TC, Magruder JT, Grimm JC, Suarez-Pierre A, Sciortino CM, Mandal K, Zehr KJ, Conte JV, Higgins RS, Cameron DE, Whitman GJ. Complications After Cardiac Operations: All Are Not Created Equal. Ann Thorac Surg. 2017 Jan;103(1):32-40. doi: 10.1016/j.athoracsur.2016.10.022. Epub 2016 Nov 22. PMID 27884410
- [Result] Echahidi N, Pibarot P, O'Hara G, Mathieu P. Mechanisms, prevention, and treatment of atrial fibrillation after cardiac surgery. J Am Coll Cardiol. 2008 Feb 26;51(8):793-801. doi: 10.1016/j.jacc.2007.10.043. PMID 18294562
- [Result] Gudbjartsson T, Helgadottir S, Sigurdsson MI, Taha A, Jeppsson A, Christensen TD, Riber LPS. New-onset postoperative atrial fibrillation after heart surgery. Acta Anaesthesiol Scand. 2020 Feb;64(2):145-155. doi: 10.1111/aas.13507. Epub 2019 Dec 2. PMID 31724159
- [Result] Melduni RM, Koshino Y, Shen WK. Management of arrhythmias in the perioperative setting. Clin Geriatr Med. 2012 Nov;28(4):729-43. doi: 10.1016/j.cger.2012.08.006. PMID 23101581
- [Result] Lopes LA, Agrawal DK. Post-Operative Atrial Fibrillation: Current Treatments and Etiologies for a Persistent Surgical Complication. J Surg Res (Houst). 2022;5(1):159-172. doi: 10.26502/jsr.10020209. Epub 2022 Mar 28. PMID 35445200